CLINICAL TRIAL: NCT00331773
Title: A Phase III Randomized Study of Hypofractionated 3D-CRT/MRT Versus Conventionally Fractionated 3D-CRT/MRT in Patients With Favorable-Risk Prostate Cancer
Brief Title: Radiation Therapy in Treating Patients With Stage II Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-0415; CDR0000481119; NCI-2009-00721 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2006-05-30; First posted 2006-05-31 (Estimated); Results first posted 2017-04-13 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2022-12

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IIB prostate cancer; stage IIA prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy, Intensity-Modulated; Radiotherapy, Conformal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional 3D-CRT (Active Comparator): Conventional 3D-CRT or IMRT to 73.8 Gy in 41 fractions
  Interventions: Radiation: Conventional 3D-CRT or IMRT
- Hypofractionated 3D-CRT (Experimental): Hypofractionated 3D-CRT or IMRT to 70 Gy in 28 fractions
  Interventions: Radiation: Hypofractionated 3D-CRT or IMRT

INTERVENTIONS:
Radiation: Conventional 3D-CRT or IMRT — Radiation therapy will be given once daily, five days a week, at 1.8 Gy per fraction, for 41 fractions and a total dose of 73.8 Gy
  Other Names: 3-dimensional conformal radiation therapy; Intensity-modulated radiation therapy (IMRT)
  Arms: Conventional 3D-CRT
Radiation: Hypofractionated 3D-CRT or IMRT — Radiation therapy will be given once daily, five days a week, at 2.5 Gy per fraction, for 28 fractions and a total dose of 70 Gy.
  Other Names: Hypofractionated 3-dimensional conformal radiation therapy; Intensity-modulated radiation therapy (IMRT)
  Arms: Hypofractionated 3D-CRT

SUMMARY:
RATIONALE: Giving radiation therapy that uses a 3-dimensional (3-D) image of the tumor to help focus thin beams of radiation directly on the tumor, and giving hypofractionated radiation therapy (higher doses over a shorter period of time), may be less costly with fewer side effects and just as effective in treating prostate cancer.

PURPOSE: This randomized phase III trial is studying several different radiation therapy regimens to compare how well they work in treating patients with stage II prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the disease-free survival (DFS) of patients with favorable-risk stage II prostate cancer treated with hypofractionated vs conventionally fractionated three-dimensional conformal radiotherapy (3D-CRT) or intensity-modulated radiotherapy (IMRT).

Secondary

* Compare time to local progression, freedom from biochemical recurrence, and disease-specific and overall survival of patients treated with these regimens.
* Determine the incidence of gastrointestinal and genitourinary toxic effects in patients treated with these regimens.
* Compare the degree, duration, and significant differences in disease-specific health-related quality of life (HRQOL) decrements, using the Expanded Prostate Cancer Index Composite (EPIC), in patients treated with these regimens.
* Determine whether anxiety and/or depression, as measured by the Hopkins Symptom Checklist-25 (HSCL-25), are decreased with therapy that improves DFS of these patients .
* Determine whether the incremental gain in DFS outweighs decrements in the generic domains of HRQOL (i.e., mobility, self care, usual activities, pain/discomfort, and anxiety/depression) in patients treated with these regimens.
* Conduct a cost-utility analysis of hypofractionated 3D-CRT or IMRT as a prostate cancer therapy if this regimen is shown to be as effective as conventionally fractionated 3D-CRT or IMRT in improving DFS.

OUTLINE: This is a randomized, controlled, multicenter study. Patients are stratified according to Gleason score (2-4 vs 5-6), prostate-specific antigen (PSA) level (< 4 ng/mL vs 4-<9 ng/mL), and planned radiotherapy modality (three-dimensional conformal radiotherapy [3D-CRT] vs intensity-modulated radiotherapy [IMRT]). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo conventionally fractionated 3D-CRT or IMRT once daily 5 days a week for 8.2 weeks (total of 41 treatments).
* Arm II: Patients undergo hypofractionated 3D-CRT or IMRT once daily 5 days a week for 5.6 weeks (total of 28 treatments).

Quality of life, anxiety, and depression are assessed at baseline and then at 6 months and 1, 2, and 5 years after the start of radiotherapy.

After completion of study treatment, patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 1,067 patients will be accrued to this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate within the past 6 months

  * Clinical stage T1-2c
* Combined Gleason score 2-6
* Prostate-specific antigen (PSA) < 10 ng/mL within the past 6 months

  * PSA evaluated at least 10 days after prostate biopsy
  * For patients who received finasteride, PSA evaluated at least 30 after completion of finasteride
  * For patients who received dutasteride, PSA evaluated at least 90 after completion of dutasteride
* No regional lymph node involvement
* No distant metastases

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-1
* No unstable angina and/or congestive heart failure requiring hospitalization within the past 6 months
* No transmural myocardial infarction within the past 6 months
* No acute bacterial or fungal infection requiring IV antibiotics
* No chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study treatment
* No hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
* No known AIDS
* No prior or concurrent lymphomatous/hematogenous malignancy or other invasive malignancy except nonmelanomatous skin cancer or any other cancer for which the patient has been continually disease-free for ≥ 5 years (e.g., carcinoma in situ of the bladder or oral cavity)
* No other severe, active comorbidity

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior radical prostatectomy or cryosurgery for prostate cancer
* No prior hormonal therapy, including any of the following:

  * Luteinizing hormone-releasing hormone agonists (e.g., goserelin or leuprolide)
  * Antiandrogens (e.g., flutamide or bicalutamide)
  * Estrogens [e.g., diethylstilbestrol (DES)]
  * Surgical castration (bilateral orchiectomy)
* No prior pelvic radiotherapy or prostate brachytherapy
* No prior or concurrent cytotoxic chemotherapy for prostate cancer
* At least 30 days since prior finasteride
* At least 90 days since prior dutasteride
* No concurrent neoadjuvant or adjuvant hormonal therapy
* Concurrent warfarin or other blood-thinning agents allowed

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1116 (Actual)
Dates: Start 2006-04 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2022-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: W. Robert Lee, MD, MS, Principal Investigator — Duke Cancer Institute; Mahul B Amin, MD, Study Chair — Cedars-Sinai Medical Center; Deborah W Bruner, RN, PhD, Study Chair — University of Pennsylvania; Daniel Low, PhD, Study Chair — Washington University School of Medicine; Gregory P Swanson, MD, Study Chair — UTHSC San Antonio
Locations (296):
- United States (282):
  - Arizona Oncology Services Foundation, Phoenix, Arizona
  - Arizona Oncology - Tucson, Tucson, Arizona
  - Auburn Radiation Oncology, Auburn, California
  - Alta Bates Summit Comprehensive Cancer Center, Berkeley, California
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - Peninsula Medical Center, Burlingame, California
  - Radiation Oncology Centers - Cameron Park, Cameron Park, California
  - Mercy Cancer Center at Mercy San Juan Medical Center, Carmichael, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Valley Medical Oncology Consultants - Castro Valley, Castro Valley, California
  - Valley Medical Oncology, Fremont, California
  - Marin Cancer Institute at Marin General Hospital, Greenbrae, California
  - Sutter Health - Western Division Cancer Research Group, Greenbrae, California
  - Kaiser Permanente Medical Center - Hayward, Hayward, California
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - Kaiser Permanente Medical Center - Los Angeles, Los Angeles, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Breast Surgeons, Incorporated, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Larry G Strieff MD Medical Corporation, Oakland, California
  - Tom K Lee, Incorporated, Oakland, California
  - Kaiser Permanente - Division of Research - Oakland, Oakland, California
  - Kaiser Permanente Medical Center - Oakland, Oakland, California
  - Valley Medical Oncology Consultants - Pleasanton, Pleasanton, California
  - Kaiser Permanente Medical Center - Rancho Cordova, Rancho Cordova, California
  - Kaiser Permanente Medical Center - Redwood City, Redwood City, California
  - Kaiser Permanente Medical Center - Richmond, Richmond, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente Medical Center - Roseville, Roseville, California
  - Radiation Oncology Center - Roseville, Roseville, California
  - Radiological Associates of Sacramento Medical Group, Incorporated, Sacramento, California
  - University of California Davis Cancer Center, Sacramento, California
  - Mercy General Hospital, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - South Sacramento Kaiser-Permanente Medical Center, Sacramento, California
  - Kaiser Permanente Medical Center - Sacramento, Sacramento, California
  - Kaiser Permanente Medical Center - San Francisco Geary Campus, San Francisco, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - California Pacific Medical Center - California Campus, San Francisco, California
  - Kaiser Permanente Medical Center - Santa Teresa, San Jose, California
  - Doctors Medical Center - San Pablo Campus, San Pablo, California
  - Kaiser Foundation Hospital - San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara Kiely Campus, Santa Clara, California
  - Santa Clara, California
  - Kaiser Permanente Medical Center - Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Medical Center - South San Francisco, South San Francisco, California
  - Kaiser Permanente Medical Facility - Stockton, Stockton, California
  - General Robert Huyser Cancer Center at David Grant Medical Center, Travis Air Force Base, California
  - Solano Radiation Oncology Center, Vacaville, California
  - Sutter Solano Medical Center, Vallejo, California
  - Kaiser Permanente Medical Center - Walnut Creek, Walnut Creek, California
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Rocky Mountain Cancer Centers - Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Radiation Oncology, Fort Collins, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Baptist-South Miami Regional Cancer Program, Miami, Florida
  - Bay Medical, Panama City, Florida
  - Georgia Cancer Center for Excellence at Grady Memorial Hospital, Atlanta, Georgia
  - Emory Crawford Long Hospital, Atlanta, Georgia
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Saint James Hospital and Health Centers Comprehensive Cancer Institute - Olympia Fields, Olympia Fields, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Methodist Cancer Center at Methodist Hospital, Indianapolis, Indiana
  - Central Indiana Cancer Centers - East, Indianapolis, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Kansas City Cancer Centers - Southwest, Overland Park, Kansas
  - Norton Suburban Hospital, Louisville, Kentucky
  - James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Central Maryland Oncology Center, Columbia, Maryland
  - Tate Cancer Center at Baltimore Washington Medical Center, Glen Burnie, Maryland
  - Helen P. Denit Cancer Center at Montgomery General Hospital, Olney, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Hudner Oncology Center at Saint Anne's Hospital - Fall River, Fall River, Massachusetts
  - MetroWest Medical Center - Framingham Union Hospital, Framingham, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Great Lakes Cancer Institute at McLaren Regional Medical Center, Flint, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Albert Lea Cancer Center at Albert Lea Medical Center, Albert Lea, Minnesota
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - St. Luke's Hospital Cancer Care Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Immanuel St. Joseph's, Mankato, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Barnes-Jewish St. Peters Hospital - St. Peters, City of Saint Peters, Missouri
  - St. John's Regional Medical Center, Joplin, Missouri
  - Kansas City Cancer Centers - South, Kansas City, Missouri
  - Kansas City Cancer Centers - North, Kansas City, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates - Reno, Reno, Nevada
  - Dartmouth - Hitchcock Concord, Concord, New Hampshire
  - Center for Cancer Care at Exeter Hospital, Exeter, New Hampshire
  - Kingsbury Center for Cancer Care at Cheshire Medical Center, Keene, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cancer Institute of New Jersey at Cooper University Hospital - Camden, Camden, New Jersey
  - CentraState Medical Center, Freehold, New Jersey
  - Princeton Radiation Oncology Center, Jamesburg, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - University Medical Center at Princeton, Princeton, New Jersey
  - Frederick R. and Betty M. Smith Cancer Treatment Center, Sparta, New Jersey
  - Capital Health Regional Cancer Center, Trenton, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua West Jersey, Voorhees Township, New Jersey
  - Lovelace Medical Center - Downtown, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New York Oncology Hematology, PC at Albany Regional Cancer Care, Albany, New York
  - Lourdes Regional Cancer Center, Binghamton, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - Cayuga Medical Center of Ithaca, Ithaca, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Don Monti Comprehensive Cancer Center at North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - Hudson Valley Oncology Associates, Poughkeepsie, New York
  - Saint Francis Hospital Cancer Center, Poughkeepsie, New York
  - Highland Hospital of Rochester, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CaroMont Cancer Center at Gaston Memorial Hospital, Gastonia, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Barberton Citizens Hospital, Barberton, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Cleveland Clinic Cancer Center at Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center, Independence, Ohio
  - Hillcrest Cancer Center at Hillcrest Hospital, Mayfield Heights, Ohio
  - Cancer Care Center, Incorporated, Salem, Ohio
  - Precision Radiotherapy at University Pointe, West Chester, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Willamette Valley Cancer Center - Eugene, Eugene, Oregon
  - Celilo Cancer Center at Mid-Columbia Medical Center, The Dalles, Oregon
  - Rosenfeld Cancer Center at Abington Memorial Hospital, Abington, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Mercy Fitzgerald Hospital, Darby, Pennsylvania
  - Northeast Radiation Oncology Center, Dunmore, Pennsylvania
  - St. Mary Regional Cancer Center, Langhorne, Pennsylvania
  - Upper Delaware Valley Cancer Center, Milford, Pennsylvania
  - Cancer Center of Paoli Memorial Hospital, Paoli, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Frankford Hospital Cancer Center - Torresdale Campus, Philadelphia, Pennsylvania
  - MNAP Oncologic Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center CCOP Research Base, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - Guthrie Cancer Center at Guthrie Clinic Sayre, Sayre, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - CCOP - Main Line Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - York Cancer Center at Apple Hill Medical Center, York, Pennsylvania
  - Carolina Regional Cancer Center, Myrtle Beach, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Texas Oncology, PA at Harris Center HEB, Bedford, Texas
  - St. Joseph Regional Cancer Center, Bryan, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Texas Oncology, PA at Texas Cancer Center Dallas Southwest, Dallas, Texas
  - Klabzuba Cancer Center at Harris Methodist Fort Worth Hospital, Fort Worth, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Cancer Therapy and Research Center, San Antonio, Texas
  - Texas Oncology, PA at Texas Cancer Center - Sherman, Sherman, Texas
  - Texas Oncology, PA at Texas Oncology Cancer Center Sugar Land, Sugar Land, Texas
  - Sandra L. Maxwell Cancer Center, Cedar City, Utah
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Community Cancer Center at Rutland Regional Medical Center, Rutland, Vermont
  - Norris Cotton Cancer Center - North, Saint Johnsbury, Vermont
  - INOVA Alexandria Hospital, Alexandria, Virginia
  - Danville Regional Medical Center, Danville, Virginia
  - Sentara Cancer Institute at Sentara Norfolk General Hospital, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Veterans Affairs Medical Center - Richmond, Richmond, Virginia
  - Harrison Medical Center, Bremerton, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - Franciscan Cancer Center at St. Joseph Medical Center, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington
  - West Virginia University Health Sciences Center - Charleston, Charleston, West Virginia
  - Theda Care Cancer Institute, Appleton, Wisconsin
  - Franciscan Skemp Healthcare - La Crosse Campus, La Crosse, Wisconsin
  - Community Memorial Hospital Cancer Care Center, Menomonee Falls, Wisconsin
  - Columbia Saint Mary's Hospital - Ozaukee, Mequon, Wisconsin
  - Columbia-Saint Mary's Cancer Care Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee, Milwaukee, Wisconsin
  - All Saints Cancer Center at Wheaton Franciscan Healthcare, Racine, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming
- Canada (14):
  - British Columbia Cancer Agency - Centre for the Southern Interior, Kelowna, British Columbia
  - BCCA - Fraser Valley Cancer Centre, Surrey, British Columbia
  - British Columbia Cancer Agency - Vancouver Cancer Centre, Vancouver, British Columbia
  - British Columbia Cancer Agency - Vancouver Island Centre, Victoria, British Columbia
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - London Regional Cancer Program at London Health Sciences Centre, London, Ontario
  - Cancer Care Program at Thunder Bay Regional Health Sciences, Thunder Bay, Ontario
  - Hopital Notre-Dame du CHUM, Montreal, Quebec
  - McGill Cancer Centre at McGill University, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan
  - Saskatoon Cancer Centre at the University of Saskatchewan, Saskatoon, Saskatchewan

REFERENCES:
- [Result] Lee WR, Dignam JJ, Amin MB, Bruner DW, Low D, Swanson GP, Shah AB, D'Souza DP, Michalski JM, Dayes IS, Seaward SA, Hall WA, Nguyen PL, Pisansky TM, Faria SL, Chen Y, Koontz BF, Paulus R, Sandler HM. Randomized Phase III Noninferiority Study Comparing Two Radiotherapy Fractionation Schedules in Patients With Low-Risk Prostate Cancer. J Clin Oncol. 2016 Jul 10;34(20):2325-32. doi: 10.1200/JCO.2016.67.0448. Epub 2016 Apr 4. PMID 27044935
- [Derived] Lee WR, Dignam JJ, Amin MB, Bruner DW, Low D, Swanson GP, Shah AB, D'Souza D, Michalski JM, Dayes IS, Seaward SA, Hall WA, Nguyen PL, Pisansky TM, Faria SL, Chen Y, Rodgers JP, Sandler HM. Long-Term Analysis of NRG Oncology RTOG 0415: A Randomized Phase III Noninferiority Study Comparing Two Fractionation Schedules in Patients With Low-Risk Prostate Cancer. J Clin Oncol. 2024 Jul 10;42(20):2377-2381. doi: 10.1200/JCO.23.02445. Epub 2024 May 17. PMID 38759121
- [Derived] Alexander GS, Krc RF, Assif JW, Sun K, Molitoris JK, Tran P, Rana Z, Bentzen SM, Mishra MV. Conditional Risks of Biochemical Failure and Prostate Cancer-Specific Death in Patients Undergoing External Beam Radiotherapy: A Secondary Analysis of 2 Randomized Clinical Trials. JAMA Netw Open. 2023 Sep 5;6(9):e2335069. doi: 10.1001/jamanetworkopen.2023.35069. PMID 37751207
- [Derived] Kim S, Kong JH, Lee Y, Lee JY, Kang TW, Kong TH, Kim MH, You SH. Dose-escalated radiotherapy for clinically localized and locally advanced prostate cancer. Cochrane Database Syst Rev. 2023 Mar 8;3(3):CD012817. doi: 10.1002/14651858.CD012817.pub2. PMID 36884035
- [Derived] Bai J, Pugh SL, Eldridge R, Yeager KA, Zhang Q, Lee WR, Shah AB, Dayes IS, D'Souza DP, Michalski JM, Efstathiou JA, Longo JM, Pisansky TM, Maier JM, Faria SL, Desai AB, Seaward SA, Sandler HM, Cooley ME, Bruner DW. Neighborhood Deprivation and Rurality Associated With Patient-Reported Outcomes and Survival in Men With Prostate Cancer in NRG Oncology RTOG 0415. Int J Radiat Oncol Biol Phys. 2023 May 1;116(1):39-49. doi: 10.1016/j.ijrobp.2023.01.035. Epub 2023 Feb 2. PMID 36736921
- [Derived] Khairnar R, DeMora L, Sandler HM, Lee WR, Villalonga-Olives E, Mullins CD, Palumbo FB, Bruner DW, Shaya FT, Bentzen SM, Shah AB, Malone S, Michalski JM, Dayes IS, Seaward SA, Albert M, Currey AD, Pisansky TM, Chen Y, Horwitz EM, DeNittis AS, Feng F, Mishra MV. Methodological Comparison of Mapping the Expanded Prostate Cancer Index Composite to EuroQoL-5D-3L Using Cross-Sectional and Longitudinal Data: Secondary Analysis of NRG/RTOG 0415. JCO Clin Cancer Inform. 2022 Jun;6:e2100188. doi: 10.1200/CCI.21.00188. PMID 35776901
- [Derived] Bruner DW, Pugh SL, Lee WR, Hall WA, Dignam JJ, Low D, Swanson GP, Shah AB, Malone S, Michalski JM, Dayes IS, Seaward SA, Nguyen PL, Pisansky TM, Chen Y, Sandler HM, Movsas B. Quality of Life in Patients With Low-Risk Prostate Cancer Treated With Hypofractionated vs Conventional Radiotherapy: A Phase 3 Randomized Clinical Trial. JAMA Oncol. 2019 May 1;5(5):664-670. doi: 10.1001/jamaoncol.2018.6752. PMID 30763425
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Groups:
- Conventional 3D-CRT: Conventional 3D-CRT or intensity-modulated radiotherapy (IMRT): Radiation therapy will be given once daily, five days a week, at 1.8 Gy per fraction, for 41 fractions and a total dose of 73.8 Gy
Period: Overall Study
Arm/Group | Conventional 3D-CRT | Hypofractionated 3D-CRT
Started | 558 | 557
Completed | 542 (Subjects with data available for the primary analysis are considered to have completed the study.) | 550 (Subjects with data available for the primary analysis are considered to have completed the study.)
Not Completed | 16 | 7
Not completed — Withdrawal by Subject | 6 | 4
Not completed — Protocol Violation | 10 | 3

BASELINE CHARACTERISTICS:
Population: Eligible patients who did not withdraw consent.
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional 3D-CRT | Hypofractionated 3D-CRT | Total
Number analyzed (Participants) | 542 | 550 | 1092
Age, Continuous [Median (Full Range); unit: years] | 67 [42 to 85] | 67 [45 to 84] | 67 [42 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 542 | 550 | 1092

OUTCOME MEASURES:

1. Primary Outcome: Five-year Disease-free Survival (DFS) Rate
Description: Five-year rates are estimated by the Kaplan-Meier method. DFS events included local progression, distant metastatic progression, biochemical recurrence as defined by the Radiation Therapy Oncology Group (RTOG) Phoenix definition, or death from any cause. Patients who experienced second primary cancers remained under observation for DFS events.
Time Frame: Analysis occurs after all patients have been followed for five years.
Population: Eligible patients who did not withdraw consent
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Conventional 3D-CRT | Hypofractionated 3D-CRT
Number analyzed (Participants) | 542 | 550
percentage of participants | 85.3 [81.9 to 88.1] | 86.3 [83.1 to 89]
Statistical Analysis 1: Comparison: Conventional 3D-CRT vs Hypofractionated 3D-CRT; Test type: Non-Inferiority or Equivalence — This trial was designed to establish with 90% power and a two-sided significance level of 0.05 that Arm 2 (Hypofractionated 3D-CRT) results in a 5-year DFS that is not lower than Arm 1 by more than 7.65% (hazard ratio [HR] , 1.52). Patients analyzed according to assignment, with time-to event duration originating at random assignment. DFS distributions calculated using the Kaplan-Meier method. Treatment efficacy for DFS was tested by comparing cause-specific hazards with the log-rank statistic; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.64 to 1.14] — Reference arm = Conventional 3D-CRT

2. Secondary Outcome: Five-year Local Progression Rate
Description: Clinical criteria for local recurrence are progression (increase in palpable abnormality) at any time, failure of regression of the palpable tumor by 2 years, and redevelopment of a palpable abnormality after complete disappearance of previous abnormalities. Histologic criteria for local recurrence are presence of prostatic carcinoma upon biopsy and positive biopsy of the palpably normal prostate more than 2 years after the start of treatment. The arms were not statistically compared because of an insufficient number of events.
Time Frame: Analysis occurs after all patients have been followed for five years.
Population: All eligible patients.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Conventional 3D-CRT | Hypofractionated 3D-CRT
Number analyzed (Participants) | 542 | 550
percentage of participants | 1.2 [0.5 to 2.4] | 0.4 [0.1 to 1.3]

3. Secondary Outcome: Five-year Disease-specific Survival Rate
Description: An event was death in association with any of the following conditions:
  * Primary cause of death certified as due to prostate cancer
  * Further clinical tumor progression occurring after initiation of "salvage" anti-tumor (e.g., (androgen suppression) therapy
  * A rise (that exceeds 1.0 ng/mL) in the serum prostate-specific antigen (PSA) level on at least two consecutive occasions that occurs during or after "salvage" androgen suppression therapy
  * Disease progression in the absence of any anti-tumor therapy
  * Death from a complication of therapy, irrespective of disease status. The arms were not statistically compared because of an insufficient number of events.
Time Frame: Analysis occurs after all patients have been followed for five years.
Population: All eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Conventional 3D-CRT | Hypofractionated 3D-CRT
Number analyzed (Participants) | 542 | 550
percentage of participants | 0.2 [0.0 to 1.0] | 0.2 [0.1 to 1.1]

4. Secondary Outcome: Five-year PSA Failure Rate
Description: Five-year rates are shown (cumulative incidence estimates). Note, although the protocol calls this endpoint "Freedom from biochemical recurrence", it defines the endpoint as "The time to PSA failure". An event for PSA, i.e. biochemical, failure was the first of the following: initiation of non-protocol (e.g., salvage) hormone therapy, or an increase in PSA of at least 2 ng/mL. Time to biochemical failure was measured from study entry until the date of failure.
Time Frame: Analysis occurs after all patients have been followed for five years.
Population: Eligible patients who did not withdraw consent.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Conventional 3D-CRT | Hypofractionated 3D-CRT
Number analyzed (Participants) | 542 | 550
percentage of participants | 8.1 [5.9 to 10.6] | 6.3 [4.5 to 8.6]
Statistical Analysis 1: Comparison: Conventional 3D-CRT vs Hypofractionated 3D-CRT; Test type: Non-Inferiority or Equivalence — Patients who died without biochemical failure were considered as competing risk at the time of death. Patients alive without biochemical failure at last follow-up were censored at that date. Estimates were calculated using cumulative risk and non-inferiority was assessed against a HR of 1.67. The log-rank test was used with a two-sided p-value of 0.05; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.51 to 1.17] — Reference arm = Conventional 3D-CRT

5. Secondary Outcome: Five-year Overall Survival Rate
Description: Five-year rates Kaplan-Meier estimates. Overall survival (OS) was measured from study entry until the date of death. Patients still alive at the time of analysis were censored at the date of last follow-up
Time Frame: Analysis occurs after all patients have been followed for five years.
Population: Eligible patients who did not withdraw consent.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Conventional 3D-CRT | Hypofractionated 3D-CRT
Number analyzed (Participants) | 542 | 550
percentage of participants | 93.2 [90.7 to 95.1] | 92.5 [89.9 to 94.5]
Statistical Analysis 1: Comparison: Conventional 3D-CRT vs Hypofractionated 3D-CRT; Test type: Non-Inferiority or Equivalence — Non-inferiority was assessed against a HR of 1.54, translated from a 5% difference in overall survival with 90% overall survival in the Conventional 3D-CRT arm. The log-rank test was used with a two-sided p-value of 0.05; p = 0.008, Log Rank; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.64 to 1.41] — Reference arm = Conventional 3D-CRT

6. Secondary Outcome: Frequency of Patients With GU and GI Acute and Late Toxicity
Description: The frequency of genitourinary (GU) and gastrointestinal (GI) adverse events as defined and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (version 3) were compared between treatment arms. Acute toxicity was defined as any toxicity beginning within 90 days of completion of RT, and late toxicity was defined as any toxicity beginning more than 90 days after the completion of RT. Acute and late GU and GI toxicity rates were tabulated and reported in two ways: dichotomized as < grade 2 vs ≥ grade 2, and dichotomized as < grade 3 vs ≥ grade 3. Higher grade indicates more severity.
Time Frame: Acute toxicity is measured from start of treatment to 90 days from the completion of treatment. Late toxicity is defined as toxicity occuring after 90 days from completion of treatment. Analysis occured at the time of the primary endpoint analysis.
Population: All eligible patients who started study treatment and did not withdraw consent
Measure: Number; unit: participants
Arm/Group | Conventional 3D-CRT | Hypofractionated 3D-CRT
Number analyzed (Participants) | 534 | 545
participants
  Acute GI: Grade >= 2: | 55 | 58
  Acute GI: Grade >= 3 | 3 | 4
  Acute GU: Grade >= 2 | 145 | 147
  Acute GU: Grade >= 3 | 13 | 18
  Late GI: Grade >= 2 | 75 | 121
  Late GI: Grade >= 3 | 14 | 22
  Late GU: Grade >= 2 | 121 | 161
  Late GU: Grade >= 3 | 12 | 19
Statistical Analysis 1: Comparison: Conventional 3D-CRT vs Hypofractionated 3D-CRT; Acute GI toxicity rates were tabulated and dichotomized as < grade 2 vs ≥ grade 2. To evaluate the differences by treatment arm, 2 X 2 subtables were formed and relative risk (RR) estimates with 95% confidence intervals (CIs) were computed; Test type: Superiority or Other; p = 0.85, Regression, Logistic — 2-sided; Risk Ratio (RR) = 1.03, 95% CI 2-sided [0.73 to 1.46] — Reference arm = Conventional 3D-CRT
Statistical Analysis 2: Comparison: Conventional 3D-CRT vs Hypofractionated 3D-CRT; Acute GI toxicity rates were tabulated and dichotomized as < grade 3 vs ≥ grade 3. To evaluate the differences by treatment arm, 2 X 2 subtables were formed and relative risk (RR) estimates with 95% CIs were computed; Test type: Superiority or Other; p = 0.72, Regression, Logistic — 2-sided; Risk Ratio (RR) = 1.31, 95% CI 2-sided [0.29 to 5.81] — Reference arm = Conventional 3D-CRT
Statistical Analysis 3: Comparison: Conventional 3D-CRT vs Hypofractionated 3D-CRT; Acute GU toxicity rates were tabulated and dichotomized as < grade 2 vs ≥ grade 2. To evaluate the differences by treatment arm, 2 X 2 subtables were formed and relative risk (RR) estimates with 95% CIs were computed; Test type: Superiority or Other; p = 0.95, Regression, Logistic — 2-sided; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.82 to 1.21] — Reference Arm = Conventional 3D-CRT
Statistical Analysis 4: Comparison: Conventional 3D-CRT vs Hypofractionated 3D-CRT; Acute GU toxicity rates were tabulated and dichotomized as < grade 3 vs ≥ grade 3. To evaluate the differences by treatment arm, 2 X 2 subtables were formed and relative risk (RR) estimates with 95% CIs were computed; Test type: Superiority or Other; p = 0.39, Regression, Logistic — 2-sided; Risk Ratio (RR) = 1.36, 95% CI 2-sided [0.67 to 2.74] — Reference arm = Conventional 3D-CRT
Statistical Analysis 5: Comparison: Conventional 3D-CRT vs Hypofractionated 3D-CRT; Late GI toxicity rates were tabulated and dichotomized as < grade 2 vs ≥ grade 2. To evaluate the differences by treatment arm, 2 X 2 subtables were formed and relative risk (RR) estimates with 95% CIs were computed; Test type: Superiority or Other; p = 0.005, Regression, Logistic — 2-sided; Risk Ratio (RR) = 1.59, 95% CI 2-sided [1.22 to 2.06] — Reference arm = Conventional 3D-CRT
Statistical Analysis 6: Comparison: Conventional 3D-CRT vs Hypofractionated 3D-CRT; Late GI toxicity rates were tabulated and dichotomized as < grade 3 vs ≥ grade 3. To evaluate the differences by treatment arm, 2 X 2 subtables were formed and relative risk (RR) estimates with 95% CIs were computed; Test type: Superiority or Other; p = 0.19, Regression, Logistic — 2-sided; Risk Ratio (RR) = 1.55, 95% CI 2-sided [0.80 to 2.99] — Reference arm = Conventional 3D-CRT
Statistical Analysis 7: Comparison: Conventional 3D-CRT vs Hypofractionated 3D-CRT; Late GU toxicity rates were tabulated and dichotomized as < grade 2 vs ≥ grade 2. To evaluate the differences by treatment arm, 2 X 2 subtables were formed and relative risk (RR) estimates with 95% CIs were computed; Test type: Superiority or Other; p = 0.009, Regression, Logistic — 2-sided; Risk Ratio (RR) = 1.31, 95% CI 2-sided [1.07 to 1.61] — Reference arm = Conventional 3D-CRT
Statistical Analysis 8: Comparison: Conventional 3D-CRT vs Hypofractionated 3D-CRT; Late GU toxicity rates were tabulated and dichotomized as < grade 3 vs ≥ grade 3. To evaluate the differences by treatment arm, 2 X 2 subtables were formed and relative risk (RR) estimates with 95% CIs were computed; Test type: Superiority or Other; p = 0.22, Regression, Logistic — 2-sided; Risk Ratio (RR) = 1.56, 95% CI 2-sided [0.76 to 3.18] — Reference arm = Conventional 3D-CRT

7. Secondary Outcome: Comparison of Disease-specific HRQOL Change in Expanded Prostate Cancer Index Composite (EPIC); the Utilization of Sexual Medications/Devices Supplements the EPIC
Description: Prostate cancer (PC) Health-Related Quality of Life (HRQOL) outcomes as measured by change over time in the Expanded Prostate Cancer Index Composite [EPIC], a PC HRQOL instrument measuring a broad spectrum of urinary, bowel, and sexual symptoms related to radiotherapy, is compared between arms. The EPIC questionnaire was grouped into four domains (bowel, urinary, sexual, hormonal), each with a score ranging from 0 (worst) to 100 (best), and was assessed at baseline, 6, 12, and 24 months, and 5 years. The difference in score from baseline to each time point was calculated and the Wilcoxon test statistic was used to test the null hypothesis that responses are the same across the two treatment arms vs. the alternative hypothesis that they are different, using a 2-sided alpha of 0.05 at each timepoint, resulting in an alpha of 0.0125 for each domain. Each row refers to a separate analysis.
Time Frame: Baseline, 6, 12, and 24 months, and 5 years
Population: Eligible patients with both a baseline and follow-up EPIC domain score, who did not withdraw consent
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Conventional 3D-CRT | Hypofractionated 3D-CRT
Number analyzed (Participants) | 542 | 550
units on a scale
  6 mo. EPIC Bowel Domain: number analyzed (Participants) | 371 | 401
  6 mo. EPIC Bowel Domain | -4 (12.1) | -3.7 (11.7)
  6 mo. EPIC Urinary Domain: number analyzed (Participants) | 292 | 338
  6 mo. EPIC Urinary Domain | 0 (10.5) | -1.5 (11.9)
  6 mo. EPIC Sexual Domain: number analyzed (Participants) | 274 | 310
  6 mo. EPIC Sexual Domain | -8.1 (20.9) | -7.8 (17.8)
  6 mo. EPIC Hormonal Domain: number analyzed (Participants) | 285 | 326
  6 mo. EPIC Hormonal Domain | -2.4 (10.5) | -1.8 (10)
  12 mo. EPIC Bowel Domain (n=273, 294): number analyzed (Participants) | 273 | 294
  12 mo. EPIC Bowel Domain (n=273, 294) | -3.7 (11.4) | -7.5 (14.6)
  12 mo. EPIC Urinary Domain: number analyzed (Participants) | 275 | 299
  12 mo. EPIC Urinary Domain | -0.3 (10.4) | -1.8 (13.1)
  12 mo. EPIC Sexual Domain: number analyzed (Participants) | 261 | 271
  12 mo. EPIC Sexual Domain | -8.1 (19.7) | -8.4 (20)
  12 mo. EPIC Hormonal Domain: number analyzed (Participants) | 263 | 288
  12 mo. EPIC Hormonal Domain | -1.6 (8.5) | -1.6 (9.4)
  24 mo. EPIC Bowel Domain: number analyzed (Participants) | 251 | 266
  24 mo. EPIC Bowel Domain | -4.4 (12.4) | -6 (12.7)
  24 mo. EPIC Urinary Domain: number analyzed (Participants) | 255 | 271
  24 mo. EPIC Urinary Domain | -0.5 (10.6) | -0.7 (12.4)
  24 mo. EPIC Sexual Domain: number analyzed (Participants) | 238 | 245
  24 mo. EPIC Sexual Domain | -9.7 (21.1) | -10.4 (21)
  24 mo. EPIC Hormonal Domain: number analyzed (Participants) | 244 | 253
  24 mo. EPIC Hormonal Domain | -2.4 (9.5) | -1.7 (10.5)
  60 mo. EPIC Bowel Domain: number analyzed (Participants) | 217 | 239
  60 mo. EPIC Bowel Domain | -3.6 (11.8) | -5.2 (12.6)
  60 mo. EPIC Urinary Domain: number analyzed (Participants) | 222 | 238
  60 mo. EPIC Urinary Domain | -1.2 (12.4) | -3.1 (15)
  60 mo. EPIC Sexual Domain: number analyzed (Participants) | 199 | 217
  60 mo. EPIC Sexual Domain | -13.5 (22.1) | -15.7 (24.4)
  60 mo. EPIC Hormonal Domain: number analyzed (Participants) | 209 | 226
  60 mo. EPIC Hormonal Domain | -2.1 (10.3) | -2.1 (10.4)
Statistical Analysis 1: Comparison: Conventional 3D-CRT vs Hypofractionated 3D-CRT; EPIC Bowel Domain at 6 months; Test type: Superiority or Other; p = 0.72, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Conventional 3D-CRT vs Hypofractionated 3D-CRT; EPIC Urinary Domain at 6 months; Test type: Superiority or Other; p = 0.056, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Conventional 3D-CRT vs Hypofractionated 3D-CRT; EPIC Sexual Domain at 6 months; Test type: Superiority or Other; p = 0.99, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Conventional 3D-CRT vs Hypofractionated 3D-CRT; EPIC Hormonal Domain at 6 months; Test type: Superiority or Other; p = 0.49, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Conventional 3D-CRT vs Hypofractionated 3D-CRT; EPIC Bowel Domain at 12 months; Test type: Superiority or Other; p = 0.0037, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Conventional 3D-CRT vs Hypofractionated 3D-CRT; EPIC Urinary Domain at 12 months; Test type: Superiority or Other; p = 0.062, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Conventional 3D-CRT vs Hypofractionated 3D-CRT; EPIC Sexual Domain at 12 months; Test type: Superiority or Other; p = 0.94, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Conventional 3D-CRT vs Hypofractionated 3D-CRT; EPIC Hormonal Domain at 12 months; Test type: Superiority or Other; p = 0.93, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: Conventional 3D-CRT vs Hypofractionated 3D-CRT; EPIC Bowel Domain at 24 months; Test type: Superiority or Other; p = 0.12, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: Conventional 3D-CRT vs Hypofractionated 3D-CRT; EPIC Urinary Domain at 24 months; Test type: Superiority or Other; p = 0.81, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: Conventional 3D-CRT vs Hypofractionated 3D-CRT; EPIC Sexual Domain at 24 months; Test type: Superiority or Other; p = 0.69, Wilcoxon (Mann-Whitney)
Statistical Analysis 12: Comparison: Conventional 3D-CRT vs Hypofractionated 3D-CRT; EPIC Hormonal Domain at 24 months; Test type: Superiority or Other; p = 0.68, Wilcoxon (Mann-Whitney)
Statistical Analysis 13: Comparison: Conventional 3D-CRT vs Hypofractionated 3D-CRT; EPIC Bowel Domain at 60 months; Test type: Superiority or Other; p = 0.071, Wilcoxon (Mann-Whitney)
Statistical Analysis 14: Comparison: Conventional 3D-CRT vs Hypofractionated 3D-CRT; EPIC Urinary Domain at 60 months; Test type: Superiority or Other; p = 0.047, Wilcoxon (Mann-Whitney)
Statistical Analysis 15: Comparison: Conventional 3D-CRT vs Hypofractionated 3D-CRT; EPIC Sexual Domain at 60 months; Test type: Superiority or Other; p = 0.4, Wilcoxon (Mann-Whitney)
Statistical Analysis 16: Comparison: Conventional 3D-CRT vs Hypofractionated 3D-CRT; EPIC Hormonal Domain at 60 months; Test type: Superiority or Other; p = 0.91, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: The Utilization of Sexual Medications/Devices Questionaire
Description: The Utilization of Sexual Medications/Devices questionaire is designed to assess the use of erectile aids among patients treated for prostate cancer. This instrument is used to complement the sexual symptom domain in the EPIC. The percentage of "Yes" responses to the following questions are reported: "Do you have a penile prosthesis", "Have you used an medications or devices to aid or improve erections?".
Time Frame: Baseline, 6, 12, and 24 months, and 5 years
Population: Eligible patients answering the questionaire, who did not withdraw consent
Measure: Number; unit: percentage of participants
Arm/Group | Conventional 3D-CRT | Hypofractionated 3D-CRT
Number analyzed (Participants) | 478 | 484
percentage of participants
  Baseline penile prosthesis question: number analyzed (Participants) | 399 | 414
  Baseline penile prosthesis question | 2.0 | 0.0
  Baseline medications/devices question: number analyzed (Participants) | 375 | 400
  Baseline medications/devices question | 24.5 | 23.0
  6 mo. penile prosthesis question: number analyzed (Participants) | 314 | 361
  6 mo. penile prosthesis question | 2.5 | 0.6
  6 mo. medications/devices question: number analyzed (Participants) | 292 | 345
  6 mo. medications/devices question | 25.0 | 24.1
  12 mo. penile prosthesis question: number analyzed (Participants) | 286 | 309
  12 mo. penile prosthesis question | 0.3 | 0.6
  12 mo. medications/devices question: number analyzed (Participants) | 270 | 300
  12 mo. medications/devices question | 29.6 | 30.3
  24 mo. penile prosthesis question: number analyzed (Participants) | 268 | 283
  24 mo. penile prosthesis question | 1.5 | 0
  24 mo. medications/devices question: number analyzed (Participants) | 259 | 279
  24 mo. medications/devices question | 36.3 | 33.3
  60 mo. penile prosthesis question: number analyzed (Participants) | 232 | 255
  60 mo. penile prosthesis question | 1.7 | 1.2
  60 mo. medications/devices question: number analyzed (Participants) | 227 | 252
  60 mo. medications/devices question | 35.2 | 31.7

9. Secondary Outcome: Change From Baseline in Assessment of Anxiety and Depression Using the HSCL-25
Description: Anxiety and depression were measured with the Hopkins Symptom Checklist (HSCL-25). It consists of 25 items: Part I of the HSCL-25 has 10 items for anxiety symptoms; Part II has 15 items for depression symptoms. The scale for each question includes four categories of response ("Not at all," "A little," "Quite a bit," "Extremely," rated 1 to 4, respectively). Two scores are calculated: the total score is the average of all 25 items and ranges from 0 to 100. A higher score indicates worse symptoms. The HSCL-25 tool was assessed at baseline, 6 months, 12 months, 24 months, and 5 years. For each patient, the change in score from baseline to the time point is calculated by subtracting the baseline value from the time point value.
Time Frame: Baseline, 6 months, 12 months, 24 months, and 5 years
Population: Eligible patients with a follow-up HSCL-25 who did not withdraw consent
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Conventional 3D-CRT | Hypofractionated 3D-CRT
Number analyzed (Participants) | 298 | 336
units on a scale
  6 months | 31.2 (7.8) | 31.8 (8.1)
  12 months: number analyzed (Participants) | 288 | 308
  12 months | 31.2 (7.3) | 32.2 (9)
  24 months: number analyzed (Participants) | 230 | 263
  24 months | 31.1 (7.5) | 31.7 (7.7)
  5 years: number analyzed (Participants) | 182 | 189
  5 years | 30.8 (7.1) | 32.1 (7.9)
Statistical Analysis 1: Comparison: Conventional 3D-CRT vs Hypofractionated 3D-CRT; The distribution of HSCL-25 at 6 months was calculated, and Wilcoxon test statistics were used to test the null hypothesis that responses are the same across the two treatment arms versus the alternative hypothesis that they are different. Significance level = 0.0125, two-sided test; Test type: Superiority or Other; p = 0.55, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Conventional 3D-CRT vs Hypofractionated 3D-CRT; The distribution of HSCL-25 at 12 months was calculated, and Wilcoxon test statistics were used to test the null hypothesis that responses are the same across the two treatment arms versus the alternative hypothesis that they are different. Significance level = 0.0125, two-sided test; Test type: Superiority or Other; p = 0.29, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Conventional 3D-CRT vs Hypofractionated 3D-CRT; The distribution of HSCL-25 at 24 months was calculated, and Wilcoxon test statistics were used to test the null hypothesis that responses are the same across the two treatment arms versus the alternative hypothesis that they are different. Significance level = 0.0125, two-sided test; Test type: Superiority or Other; p = 0.23, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Conventional 3D-CRT vs Hypofractionated 3D-CRT; The distribution of HSCL-25 at 60 months (5 years) was calculated, and Wilcoxon test statistics were used to test the null hypothesis that responses are the same across the two treatment arms versus the alternative hypothesis that they are different. Significance level = 0.0125, two-sided test; Test type: Superiority or Other; p = 0.028, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: EQ-5D Scores
Description: The EQ-5D is a 2-part self-assessment questionnaire. First part is 5 items (mobility, self care, usual activities, pain/discomfort, anxiety/depression) each with 3 problem levels (1-none, 2-moderate, 3-extreme). Health states are defined by the combination of the leveled responses to the 5 dimensions, generating 243 health states to which unconsciousness and death are added. The 2nd part is a visual analogue scale (VAS) valuing current health state, measured on a 20-cm 10-point interval scale. Worst imaginable health state is scored as 0 at the bottom of the scale, and best imaginable health state is scored as 100 at the top. Both the 5-item index score and the VAS score are transformed into a utility score between 0 -Worst health stat and 1 -Best health state. A two-sided Wilcoxon test with alpha 0.05 was used due to the skewed, thus non-normal, nature of the data.
Time Frame: Baseline, 6 months, 12 months, 24 months, and 5 years
Population: Eligible patients with a baseline or follow-up EQ-5D score who did not withdraw consent
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Conventional 3D-CRT | Hypofractionated 3D-CRT
Number analyzed (Participants) | 418 | 439
units on a scale
  Baseline VAS Score: number analyzed (Participants) | 402 | 430
  Baseline VAS Score | 85.0 [79.0 to 90.0] | 82.0 [75.0 to 90.0]
  Baseline Index Score: number analyzed (Participants) | 416 | 434
  Baseline Index Score | 1.0 [0.8 to 1.0] | 1.0 [0.8 to 1.0]
  6 mo. VAS Score: number analyzed (Participants) | 316 | 360
  6 mo. VAS Score | 85.0 [75.0 to 90.0] | 85.0 [75.0 to 90.0]
  6 mo. Index Score: number analyzed (Participants) | 321 | 364
  6 mo. Index Score | 1.0 [0.8 to 1.0] | 1.0 [0.8 to 1.0]
  12 mo. VAS Score: number analyzed (Participants) | 287 | 0312
  12 mo. VAS Score | 85.0 [75.0 to 90.0] | 81.5 [75.0 to 90.0]
  12 mo. Index Score: number analyzed (Participants) | 301 | 319
  12 mo. Index Score | 1.0 [0.8 to 1.0] | 1.0 [0.8 to 1.0]
  24 mo. VAS Score: number analyzed (Participants) | 276 | 280
  24 mo. VAS Score | 85.0 [75.0 to 90.0] | 85.0 [75.0 to 90.0]
  24 mo. Index Score: number analyzed (Participants) | 275 | 278
  24 mo. Index Score | 1.0 [0.8 to 1.0] | 1.0 [0.8 to 1.0]
  60 mo. VAS Score: number analyzed (Participants) | 231 | 243
  60 mo. VAS Score | 85.0 [75.0 to 90.0] | 82.0 [73.0 to 90.0]
  60 mo. Index Score: number analyzed (Participants) | 229 | 248
  60 mo. Index Score | 0.9 [0.8 to 1.0] | 0.9 [0.8 to 1.0]
Statistical Analysis 1: Comparison: Conventional 3D-CRT vs Hypofractionated 3D-CRT; Baseline VAS score; Test type: Superiority or Other; p = 0.037, Wilcoxon (Mann-Whitney); Two-sided significance level = 0.05
Statistical Analysis 2: Comparison: Conventional 3D-CRT vs Hypofractionated 3D-CRT; Baseline index score; Test type: Superiority or Other; p = 0.12, Wilcoxon (Mann-Whitney) — Two-sided significance level = 0.05
Statistical Analysis 3: Comparison: Conventional 3D-CRT vs Hypofractionated 3D-CRT; 6-month VAS score; Test type: Superiority or Other; p = 0.70, Wilcoxon (Mann-Whitney) — Two-sided significance level = 0.05
Statistical Analysis 4: Comparison: Conventional 3D-CRT vs Hypofractionated 3D-CRT; 6-month index score; Test type: Superiority or Other; p = 0.20, Wilcoxon (Mann-Whitney) — Two-sided significance level = 0.05
Statistical Analysis 5: Comparison: Conventional 3D-CRT vs Hypofractionated 3D-CRT; 12-month VAS score; Test type: Superiority or Other; p = 0.31, Wilcoxon (Mann-Whitney) — Two-sided significance level = 0.05
Statistical Analysis 6: Comparison: Conventional 3D-CRT vs Hypofractionated 3D-CRT; 12-month index score; Test type: Superiority or Other; p = 0.19, Wilcoxon (Mann-Whitney) — Two-sided significance level = 0.05
Statistical Analysis 7: Comparison: Conventional 3D-CRT vs Hypofractionated 3D-CRT; 24-month VAS score; Test type: Superiority or Other; p = 0.86, Wilcoxon (Mann-Whitney) — Two-sided significance level = 0.05
Statistical Analysis 8: Comparison: Conventional 3D-CRT vs Hypofractionated 3D-CRT; 24-month index score; Test type: Superiority or Other; p = 0.45, Wilcoxon (Mann-Whitney) — Two-sided significance level = 0.05
Statistical Analysis 9: Comparison: Conventional 3D-CRT vs Hypofractionated 3D-CRT; 60-month VAS score; Test type: Superiority or Other; p = 0.39, Wilcoxon (Mann-Whitney) — Two-sided significance level = 0.05
Statistical Analysis 10: Comparison: Conventional 3D-CRT vs Hypofractionated 3D-CRT; 60-month index score; Test type: Superiority or Other; p = 0.56, Wilcoxon (Mann-Whitney) — Two-sided significance level = 0.05

11. Secondary Outcome: Assessment of Trade-off Between Disease-free Survival and Quality of Life.
Description: To examine trade-offs between the survival time and QOL, we were to combine them for each patient into two single measurements: quality adjusted live year (QALY) and quality adjusted disease-free survival year (QADFSY). We were to use Glasziou's multiple health-state (Q-TWiST) models to use the repeated measures of EQ-5D.
Time Frame: From baseline to 5 years from the start of treatment
Population: This analysis was not conducted because there were no differences in EQ-5D scores. See results presented for Outcome Measure 10: Evaluation and Comparison of the Cost-utility of Each Treatment Arm Using EQ-5D.
Arm/Group | Conventional 3D-CRT | Hypofractionated 3D-CRT
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Statistical Modeling of Genomic Biomarkers
Time Frame: Baseline biomarker collection. Analysis would occur after the primary endpoint analysis.
Population: The protocol did not provide sufficient detail to meet National Cancer Institute requirements for release of specimens from the NRG tissue bank for the protocol-specified analysis, therefore no assays were performed and no data were collected for this outcome measure. Specimen use will require federal approval and funding separate from this trial.
Arm/Group | Conventional 3D-CRT | Hypofractionated 3D-CRT
Number analyzed (Participants) | 0 | 0

13. Other Pre Specified Outcome: Collection of Paraffin-embedded Tissue Block, Serum, Plasma, and Buffy Coat Cells for Future Translational Research Analyses
Time Frame: From baseline to 5 years from the start of treatment.
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Eligible patients with adverse event data who started study treatment are included. Patients experiencing more than one of a given adverse event are counted only once for that adverse event.
Groups:
- Conventional 3D-CRT: CConventional 3D-CRT or IMRT: Radiation therapy will be given once daily, five days a week, at 1.8 Gy per fraction, for 41 fractions and a total dose of 73.8 Gy
Arm/Group | Conventional 3D-CRT | Hypofractionated 3D-CRT
Serious Adverse Events (participants affected / at risk) | 28/534 | 32/545
Other Adverse Events (participants affected / at risk) | 466/534 | 497/545
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Conventional 3D-CRT (N=534) | Hypofractionated 3D-CRT (N=545)
Blood/bone marrow - Other (Blood and lymphatic system disorders) | 0 | 1
Hemoglobin (Blood and lymphatic system disorders) | 1 | 0
Arrhythmia NOS (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhea NOS (Gastrointestinal disorders) | 2 | 0
Duodenal obstruction (Gastrointestinal disorders) | 1 | 0
Fecal incontinence (Gastrointestinal disorders) | 1 | 0
Gastrointestinal - Other (Gastrointestinal disorders) | 1 | 0
Pancreatitis NOS (Gastrointestinal disorders) | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 1
Proctitis NOS (Gastrointestinal disorders) | 3 | 2
Rectal hemorrhage (Gastrointestinal disorders) | 2 | 2
Rectal perforation (Gastrointestinal disorders) | 1 | 0
Edema: limb (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Cholecystitis NOS (Hepatobiliary disorders) | 0 | 1
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Gallbladder (cholecystitis) (Infections and infestations) | 0 | 1
Pneumonia NOS (Infections and infestations) | 1 | 0
Hypercholesterolemia (Investigations) | 0 | 1
Metabolic/laboratory - Other (Investigations) | 1 | 0
Acidosis NOS (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness, generalized or specific area (not due to neuropathy): Extremity-lower (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Cerebral ischemia (Nervous system disorders) | 0 | 2
Convulsions NOS (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Libido decreased (Psychiatric disorders) | 1 | 0
Bladder obstruction (Renal and urinary disorders) | 0 | 1
Bladder pain (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 4 | 5
Renal/genitourinary - Other (Renal and urinary disorders) | 0 | 2
Urethral stricture (Renal and urinary disorders) | 1 | 0
Urinary bladder hemorrhage (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 2
Urinary retention (Renal and urinary disorders) | 2 | 2
Ejaculatory disorder NOS (Reproductive system and breast disorders) | 1 | 0
Erectile dysfunction NOS (Reproductive system and breast disorders) | 4 | 3
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Conventional 3D-CRT (N=534) | Hypofractionated 3D-CRT (N=545)
Constipation (Gastrointestinal disorders) | 55 | 59
Diarrhea NOS (Gastrointestinal disorders) | 173 | 211
Fecal incontinence (Gastrointestinal disorders) | 17 | 35
Gastrointestinal - Other (Gastrointestinal disorders) | 49 | 72
Hemorrhoids (Gastrointestinal disorders) | 36 | 52
Proctitis NOS (Gastrointestinal disorders) | 117 | 162
Rectal hemorrhage (Gastrointestinal disorders) | 88 | 137
Fatigue (General disorders) | 161 | 155
Pain - Other (General disorders) | 32 | 41
Libido decreased (Psychiatric disorders) | 28 | 35
Bladder pain (Renal and urinary disorders) | 31 | 25
Cystitis NOS (Renal and urinary disorders) | 88 | 107
Pollakiuria (Renal and urinary disorders) | 378 | 404
Renal/genitourinary - Other (Renal and urinary disorders) | 84 | 126
Urethral pain (Renal and urinary disorders) | 15 | 32
Urinary incontinence (Renal and urinary disorders) | 64 | 90
Urinary retention (Renal and urinary disorders) | 123 | 143
Ejaculatory disorder NOS (Reproductive system and breast disorders) | 30 | 34
Erectile dysfunction NOS (Reproductive system and breast disorders) | 199 | 214

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.